CLINICAL TRIAL: NCT02639585
Title: Efficacy and Safety of Daclatasvir Plus Asunaprevir Treatment in Patients With Chronic Hepatitis C : Prospective Cohort Study
Brief Title: Efficacy and Safety of Daclatasvir Plus Asunaprevir in Chronic Hepatitis C
Acronym: ESDAC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Won Lim, Assistant Professor, Department of Internal Medicine, Pusan National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESDAC
Record Dates: First submitted 2015-12-21; First posted 2015-12-24 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Hepatitis C, Chronic
Keywords: daclatasvir; asunaprevir
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment arm (Experimental): Daclinza and Sunvepra
  Interventions: Drug: Daclinza and Sunvepra

INTERVENTIONS:
Drug: Daclinza and Sunvepra — direct acting antiviral agent against to hepatitis C virus

SUMMARY:
We perform this study to identity efficacy and safety of Daclatasvir and Asunaprevir in real practice.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Males and females, ≥ 18 years of age
3. HCV Genotype 1b who previously failed treatment with peginterferon alfa and ribavirin, classified as previous null or partial responders based on previous therapy, OR intolerant or ineligible to P/R due to neutropenia, anemia, depression or thrombocytopenia with fibrosis/cirrhosis, OR treatment naive
4. HCV RNA ≥ 10,000 IU/mL
5. Subjects with compensated cirrhosis are permitted
6. Seronegative for Human immunodeficiency virus (HIV) and Hepatitis B surface antigen (HBsAg)
7. Negative urine or serum pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of test drug. Additionally, all fertile males with partners of childbearing age and all females with childbearing potential must use reliable contraception method during the study and for 3 months after treatment completion.

Exclusion Criteria:

1. Inability or unwillingness to provide informed consent or abide by the requirements of the study
2. Other than genotype 1 infection
3. Prior treatment of HCV with HCV direct acting antiviral agents (DAA)
4. Patient who has any history of major organ transplantation with an existing functional graft or Patient who has plan to receive organ transplant
5. Diagnosed or suspected hepatocellular carcinoma or other malignancies
6. Evidence of decompensated liver disease including, but not limited to, a history or presence of ascites, bleeding varices, or hepatic encephalopathy
7. Evidence of a medical condition contributing to chronic liver disease other than HCV
8. Uncontrolled diabetes or hypertension
9. Women with ongoing pregnancy or who are breast feeding
10. Evidence of alcohol and/or drug abuse
11. Patient who has NS5A resistance associated variant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-02 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Sustained Virologic Responase | week 12 (after treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Won Lim, M.S., Principal Investigator — Pusan National University Hospital; Young Mi Hong, M.S., Principal Investigator — Pusan National University Yangsan Hospital
Locations (2):
- South Korea (2):
  - Pusan National University Hospital, Busan
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferenci P, Bernstein D, Lalezari J, Cohen D, Luo Y, Cooper C, Tam E, Marinho RT, Tsai N, Nyberg A, Box TD, Younes Z, Enayati P, Green S, Baruch Y, Bhandari BR, Caruntu FA, Sepe T, Chulanov V, Janczewska E, Rizzardini G, Gervain J, Planas R, Moreno C, Hassanein T, Xie W, King M, Podsadecki T, Reddy KR; PEARL-III Study; PEARL-IV Study. ABT-450/r-ombitasvir and dasabuvir with or without ribavirin for HCV. N Engl J Med. 2014 May 22;370(21):1983-92. doi: 10.1056/NEJMoa1402338. Epub 2014 May 4. PMID 24795200
- [Background] Zeuzem S, Jacobson IM, Baykal T, Marinho RT, Poordad F, Bourliere M, Sulkowski MS, Wedemeyer H, Tam E, Desmond P, Jensen DM, Di Bisceglie AM, Varunok P, Hassanein T, Xiong J, Pilot-Matias T, DaSilva-Tillmann B, Larsen L, Podsadecki T, Bernstein B. Retreatment of HCV with ABT-450/r-ombitasvir and dasabuvir with ribavirin. N Engl J Med. 2014 Apr 24;370(17):1604-14. doi: 10.1056/NEJMoa1401561. Epub 2014 Apr 10. PMID 24720679
- [Background] Manns M, Pol S, Jacobson IM, Marcellin P, Gordon SC, Peng CY, Chang TT, Everson GT, Heo J, Gerken G, Yoffe B, Towner WJ, Bourliere M, Metivier S, Chu CJ, Sievert W, Bronowicki JP, Thabut D, Lee YJ, Kao JH, McPhee F, Kopit J, Mendez P, Linaberry M, Hughes E, Noviello S; HALLMARK-DUAL Study Team. All-oral daclatasvir plus asunaprevir for hepatitis C virus genotype 1b: a multinational, phase 3, multicohort study. Lancet. 2014 Nov 1;384(9954):1597-605. doi: 10.1016/S0140-6736(14)61059-X. Epub 2014 Jul 28. PMID 25078304